CLINICAL TRIAL: NCT00514514
Title: Multi-center, Open-label, Prospective, Randomized, Parallel Group, Long-term Study Investigating a Standard Regimen in de Novo Kidney Transplant Patients Versus a CNI-free Regimen and a CNI-low Dose Regimen
Brief Title: Study Investigating a Standard Regimen in de Novo Kidney Transplant Patients Versus a Calcineurin Inhibitor (CNI)-Free Regimen and a CNI-low Dose Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ADE13; 2006-007021-32
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Results first posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
Keywords: Everolimus; mycophenolate; CNI-free; kidney transplantation
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Cyclosporine; Basiliximab

ARMS (3):
- CNI standard regimen (Active Comparator): Myfortic, Sandimmun Optoral and corticosteroids
  Interventions: Drug: Myfortic; Drug: Sandimmun Optoral; Drug: Simulect®
- CNI free regimen (Experimental): CNI free regimen: comprising the following steps for switching treatment:
  Step 1 at BL2 + 1 day: Myfortic, Certican 1.5 mg, Sandimmun Optoral (50% of standard dose) and corticosteroids Step 2 at BL2 + 8 days: Myfortic, Certican 3 mg and corticosteroids
  Interventions: Drug: Everolimus; Drug: Myfortic; Drug: Sandimmun Optoral
- CNI low regimen (Active Comparator): CNI low regimen: comprising the following steps for switching treatment:
  Step 1 at BL2 + 1 day: Certican 1.5 mg, Sandimmun Optoral and corticosteroids Step 2 at BL2 + 8 days: Certican 1.5 mg, Sandimmun Optoral (low dose) and corticosteroids
  Interventions: Drug: Everolimus; Drug: Sandimmun Optoral

INTERVENTIONS:
Drug: Everolimus — Tablet containing 0.5 mg or 0.75 mg. Dosing schedule: Initially 1.5 mg/day, then based on blood level (5-10 ng/mL in CNI free, 3-8 ng/mL in CNI low regimen
  Other Names: Certican
  Arms: CNI free regimen; CNI low regimen
Drug: Myfortic — 1 tablet containing 180 mg or 360 mg
  Dosing schedule:
  Initially 1.5 mg/day, then based on blood level (5-10 ng/mL in CNI free, 3-8 ng/mL in CNI low regimen) According to blood level 1440 mg/day (2 x 720 mg), if tolerated. Dose reduction possible in case of side effects (min. dose at BL2 (Month 3): 720 mg/day)
  Other Names: Enteric Coated Mycophenolate Sodium
  Arms: CNI free regimen; CNI standard regimen
Drug: Sandimmun Optoral — 1 capsule containing 10, 25, 50, or 100mg. Dosing: According to blood level
  Other Names: Cyclosporine A
Drug: Simulect® — Lyophilisate in vials with ampoules of sterile water for injection (5 ml). Dosing: 1 vial containing 20 mg lyophilisate. Dosing schedule: 2 x 20 mg to be applied as 10 sec. bolus injection, i.v. on Day 0 (2 h before transplant) and on Day 4
  Other Names: Basiliximab
  Arms: CNI standard regimen

SUMMARY:
The purpose of this study is to compare renal function of immunosuppressive regimens with different relevance of the calcineurin inhibitor (CNI) cyclosporine: standard dose CNI, low dose CNI, CNI free in de novo kidney transplant patients after 12 months of therapy.

ELIGIBILITY:
Inclusion criteria

* Males or females, aged 18 - 70 years
* Recipients of de novo cadaveric, living unrelated or living related kidney transplants
* Females capable of becoming pregnant must have a negative serum pregnancy test within 7 days prior to or at screening, and are required to practice an approved method of birth control for the duration of the study and for a period of 6 weeks following discontinuation of study medication, even where there has been a history of infertility.
* Patients who are willing and able to participate in the study and from whom written informed consent has been obtained.

Exclusion criteria

* More than one previous renal transplantation
* Multi-organ recipients (e.g., kidney and pancreas) or previous transplant with any other organ, different from kidney
* Patients receiving a kidney from a non-heart beating donor
* Donor age: < 5 years or > 70 years
* Graft loss due to immunological reasons in the first year after transplantation (in case of secondary transplantation)
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2007-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Director — Novartis
Locations (16):
- Germany (15):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hannover Muenden
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kaiserslautern
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensburg
- Novartis Investigative Site, Bern, Switzerland

REFERENCES:
- [Derived] Sommerer C, Witzke O, Lehner F, Arns W, Reinke P, Eisenberger U, Vogt B, Heller K, Jacobi J, Guba M, Stahl R, Hauser IA, Kliem V, Wuthrich RP, Muhlfeld A, Suwelack B, Duerr M, Paulus EM, Zeier M, Porstner M, Budde K; ZEUS and HERAKLES study investigators. Onset and progression of diabetes in kidney transplant patients receiving everolimus or cyclosporine therapy: an analysis of two randomized, multicenter trials. BMC Nephrol. 2018 Sep 19;19(1):237. doi: 10.1186/s12882-018-1031-1. PMID 30231851
- [Derived] Budde K, Zeier M, Witzke O, Arns W, Lehner F, Guba M, Jacobi J, Kliem V, Reinke P, Hauser IA, Vogt B, Stahl R, Rath T, Duerr M, Paulus EM, May C, Porstner M, Sommerer C; HERAKLES Study Group. Everolimus with cyclosporine withdrawal or low-exposure cyclosporine in kidney transplantation from Month 3: a multicentre, randomized trial. Nephrol Dial Transplant. 2017 Jun 1;32(6):1060-1070. doi: 10.1093/ndt/gfx075. PMID 28605781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: .817 patients were screened and 802 were enrolled on Day of transplant which served as Baseline Visit 1. For three months post transplantation, in the pre-phase period, all patients received induction therapy (Simulect®) and immunosuppressive therapy consisting of Myfortic, Sandimmun Optoral and corticosteroids.
Pre-assignment Details: At month 3 post transplant, Baseline Visit 2, additional eligibility was assessed and patients randomized to one of 3 treatment arms and stratified according to kidney donor (living or cadaveric).
Groups:
- Standard Regimen: Myfortic, Sandimmun Optoral and corticosteroids
- CNI Free Regimen: CNI free regimen: comprising the following steps for switching treatment:
  Step 1 at BL2 + 1 day: Myfortic, everolimus 1.5 mg, Sandimmun Optoral (50% of standard dose) and corticosteroids Step 2 at BL2 + 8 days: Myfortic, everolimus 3 mg and corticosteroids
- CNI Low Regimen: CNI low regimen: comprising the following steps for switching treatment:
  Step 1 at BL2 + 1 day: everolimus 1.5 mg, Sandimmun Optoral and corticosteroids Step 2 at BL2 + 8 days: everolimus 1.5 mg, Sandimmun Optoral (low dose) and corticosteroids
Period: Pre-phase
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Started | 802 (All enrolled patients received standard regimen for 3 months) | 0 | 0
Completed | 499 | 0 | 0
Not Completed | 303 | 0 | 0
Not completed — Death | 10 | 0 | 0
Not completed — administrative problems | 2 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 0
Not completed — condition no longer requires study drug | 7 | 0 | 0
Not completed — abnormal test procedure results | 15 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — abnormal lab values | 23 | 0 | 0
Not completed — Lack of Efficacy | 35 | 0 | 0
Not completed — Adverse Event | 137 | 0 | 0
Not completed — Withdrawal by Subject | 66 | 0 | 0
Period: Randomized - 9 Month
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Started | 166 | 171 | 162
Randomized - Received Treatment | 165 | 171 | 161
Completed | 127 | 110 | 124
Not Completed | 39 | 61 | 38
Not completed — Death | 3 | 2 | 2
Not completed — Administrative problems | 1 | 1 | 2
Not completed — Withdrawal by Subject | 7 | 7 | 5
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 3 | 1
Not completed — Abnormal laboratory values | 0 | 3 | 1
Not completed — Adverse Event | 25 | 44 | 27
Period: Extension - 4 Years
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Started | 145 | 139 | 134
Non-randomized (Followed) | 95 (Patients were not randomized but continued on standard regimen and entered follow up.) | 0 | 0
Completed | 108 | 117 | 113
Not Completed | 37 | 22 | 21
Not completed — Withdrawal by Subject | 5 | 2 | 2
Not completed — Lost to Follow-up | 12 | 10 | 9
Not completed — Administrative problems | 3 | 1 | 1
Not completed — Death | 8 | 3 | 6
Not completed — Adverse Event | 9 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen | Total
Number analyzed (Participants) | 165 | 171 | 161 | 497
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.8) | 48.9 (12.5) | 48.6 (12.3) | 49.1 (12.2)
Gender [Count of Participants; unit: Participants]
  Female | 65 | 69 | 61 | 195
  Male | 100 | 102 | 100 | 302

OUTCOME MEASURES:

1. Primary Outcome: GFR Via Nankivell Method at Month 12 - CNI-Free vs Standard Regimen
Description: Demonstrate superiority of CNI-Free vs Standard Regimen in GFR using the Nankivell formula (GFR = 6.7 / Scr + BW / 4 - Surea / 2-100 / (height)² + C where where Scr is the serum creatinine concentration expressed in mmol/L, BW the body weight in kilograms, Surea the serum urea in mmol/L, height in m, and the constant C is 35 for male and 25 for female patients. The calculated GFR is expressed in mL/min per 1.73m², last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model, with treatment, center, donor type (deceased vs. living) as factors and BL2-value at V4/M3/BL2 as covariate. P-values are not adjusted
Time Frame: From randomization at BL2 (Month 3) to Month 12 post-transplant
Population: Participants analyzed differs due to different input values requested by the different formulas (Nankivell, MDRD and Cockcroft-Gault). ITT Population consisted of all patients who were randomized at Month 3 who received at least one dose of randomized treatment. The ITT population might have included patients without any data after randomization.
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 159 | 163 | 160
ml/min/1.73m² | 63.03 [60.57 to 65.49] | 68.59 [66.10 to 71.08] | 63.08 [60.62 to 65.55]
Statistical Analysis 1: Comparison: Standard Regimen vs CNI Free Regimen; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 5.56, 95% CI 2-sided [2.82 to 8.31]

2. Secondary Outcome: GFR Via Nankivell Formula at Month 12 - All Regimens
Description: Change in GFR using the Nankivell formula (GFR = 6.7 / Scr + BW / 4 - Surea / 2-100 / (height)² + C where where Scr is the serum creatinine concentration expressed in mmol/L, BW the body weight in kilograms, Surea the serum urea in mmol/L, height in m, and the constant C is 35 for male and 25 for female patients. The calculated GFR is expressed in mL/min per 1.73m², last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model, with treatment, center, donor type (deceased vs. living) as factors and BL2-value at V4/M3/BL2 as covariate.
Time Frame: From randomization at BL2 (Month 3) to Month 12 post-transplant
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 159 | 163 | 160
ml/min/1.73m² | 63.03 [60.57 to 65.49] | 68.59 [66.10 to 71.08] | 63.08 [60.62 to 65.55]

3. Secondary Outcome: GFR at Month 12 Utilizing Modification of Diet in Renal Disease (MDRD) Method
Description: Change in GFR (Modification of Diet in Renal Disease calculated using the -MDRD formulat:
  For men: GFR = 170 × (serum creatinine -0,999)×(age-0,176) x (urea nitrogen -0,17) × (albumin0,318) For women: GFR = 170 × (serum creatinine -0,999) × (age-0,176) × (urea nitrogen -0,17) x (albumin0,318) × 0.762 with urea nitrogen = urea / 2.144. ), last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model, with treatment, center, donor type (deceased vs. living) as factors and BL2-value at V4/M3/BL2 as covariate.
Time Frame: From randomization at BL2 (Month 3) to Month 12 post-transplant
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 151 | 158 | 157
ml/min/1.73m² | 50.23 [47.66 to 52.80] | 56.36 [53.77 to 58.94] | 50.24 [47.70 to 52.77]

4. Secondary Outcome: GFR at Month 12 Utilizing Cockcroft-Gault Formula
Description: Cockcroft-Gault formula: For men: GFR= ((140-age) × body weight in kg)∕(72 x serum creatinine in mg∕dl)For women: GFR= (0.85×(140-age) × body weight in kg)∕(72 x serum creatinine in mg/dl), ), last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model
Time Frame: From randomization at BL2 (Month 3) to Month 12 post-transplant
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 160 | 164 | 160
ml/min/1.73m² | 60.18 [57.33 to 63.03] | 64.87 [61.99 to 67.75] | 61.16 [58.31 to 64.02]

5. Secondary Outcome: Mean Change in Serum Creatinine From Month 3 to Month 12
Description: Change in venous blood serum creatinine. Last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model
Time Frame: From randomization at BL2 (Month 3) to Month 12 post-transplant
Population: Participants analyzed required at least one post randomization value. ITT Population consisted of all patients who were randomized at Month 3 who received at least one dose of randomized treatment. The ITT population might have included patients without any data after randomization
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 160 | 165 | 160
mg/dl | 1.66 [1.51 to 1.81] | 1.58 [1.43 to 1.73] | 1.76 [1.61 to 1.91]

6. Secondary Outcome: Efficacy Event Data From Baseline 2 (Month 3) to Month 6
Description: Efficacy events were: Biopsy-proven acute rejection (BPAR), graft loss, death, and treatment failure (defined as composite endpoint of BPAR, graft loss, death, loss to follow-up, discontinuation due to lack of efficacy or due to toxicity).
Time Frame: From Baseline 2 (Month 3) to Month 6
Population: The Intention-to-treat (ITT) Population consisted of all patients who were randomized at BL2 (Month 3), and who received at least one dose of randomized treatment. Patients were analyzed according to their assigned treatment. The ITT population might have included patients without any data after randomization.
Measure: Number; unit: Participants
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 165 | 171 | 161
Participants
  BPAR | 6 [1.51 to 1.81] | 15 [1.43 to 1.73] | 10 [1.61 to 1.91]
  Graft loss | 0 | 1 | 1
  Death | 1 | 1 | 0
  Lost to follow-up | 0 | 0 | 0
  Discontinuation due to lack of efficacy | 1 | 2 | 1
  Discontinuation due to adverse event | 8 | 26 | 13
  Therapy failure composite | 14 | 37 | 19

7. Secondary Outcome: Efficacy Event Data Baseline 2 (Month 3) to Month 12
Description: as for outcome 6
Time Frame: From Baseline 2 (Month 3) to Month 12
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 165 | 171 | 161
Participants
  BPAR | 13 [1.51 to 1.81] | 20 [1.43 to 1.73] | 13 [1.61 to 1.91]
  Graft loss | 1 | 2 | 1
  Death | 3 | 2 | 2
  Lost to follow-up | 0 | 0 | 0
  Discontinuation due to lack of efficacy | 2 | 3 | 1
  Discontinuation due to adverse event | 25 | 44 | 27
  Therapy failure composite | 34 | 58 | 35

8. Secondary Outcome: Change From BL2 (Month 3) to Month 12 in Cardiovascular Risk (Framingham Score; 10-year Cardiovascular Risk)
Description: The Framingham Score (based on LDL cholesterol level) estimates the coronary heart disease risk (%) of developing one of the following coronary heart diseases: angina pectoris, myocardial infarction, or coronary disease death, over the course of 10 years.
Time Frame: From Baseline 2 (Month 3) to Month 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent risk
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 165 | 171 | 161
Percent risk
  Baseline 1/Visit 1 (n=165,171,161) | 10.9 (8) [1.51 to 1.81] | 10.2 (7.4) [1.43 to 1.73] | 9.5 (6.9) [1.61 to 1.91]
  Baseline 2/Month 3 (n=165,171,161) | 10.3 (7.7) | 8.8 (5.9) | 9.3 (7.2)
  Month 12 (n=158,166,156) | 9.4 (6.8) | 9.1 (6.4) | 8.7 (6.8)
  Change from Baseline 2 to Month 12 (n=158,166,156) | -0.7 (5.8) | 0.4 (5.1) | -0.7 (5.4)

9. Secondary Outcome: GFR Calculated Via Nankivell Formula at Month 60
Description: as for outcome 2
Time Frame: From randomization at BL2 (Month 3) to Month 60
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 99 | 108 | 104
ml/min/1.73m² | 60.24 [57.11 to 63.38] | 66.98 [63.78 to 70.17] | 58.74 [55.58 to 61.9]

10. Secondary Outcome: GFR at Month 60 Utilizing Cockcroft-Gault Formula
Description: Cockcroft-Gault formula: For men: GFR= ((140-age) × body weight in kg)∕(72 x serum creatinine in mg∕dl) For women: GFR= (0.85×(140-age) × body weight in kg)∕(72 x serum creatinine in mg/dl), ), last observation carried forward (LOCF) was used for imputation of missing values, ANCOVA model
Time Frame: From randomization at BL2 (Month 3) to Month 60 post-transplant
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 162 | 165 | 159
ml/min/1.73m² | 55.92 [52.36 to 59.48] | 61.6 [57.99 to 65.2] | 52.91 [49.32 to 56.5]

11. Secondary Outcome: GFR at Month 60 Utilizing Modification of Diet in Renal Disease (MDRD) Method
Description: as for outcome 3
Time Frame: From randomization at BL2 (Month 3) to Month 60 post-transplant
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m²
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 152 | 159 | 156
ml/min/1.73m² | 47.56 [44.58 to 50.54] | 53.41 [50.4 to 56.42] | 44.79 [41.83 to 47.74]

12. Secondary Outcome: Mean Change in Serum Creatinine From Month 3 to Month 60
Description: as for outcome 5
Time Frame: From randomization at BL2 (Month 3) to Month 60 post-transplant
Population: Participants analyzed were previously enrolled in the core study and had at least one serum creatinine value in the extension period.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 82 | 49 | 28
mg/dl | 1.94 [1.72 to 2.15] | 1.69 [1.47 to 1.91] | 2.01 [1.79 to 2.23]

13. Secondary Outcome: Efficacy Event Data After Month 12 to Month 60
Description: as for outcome 6
Time Frame: Events starting after Month 12
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Standard Regimen | CNI Free Regimen | CNI Low Regimen
Number analyzed (Participants) | 165 | 171 | 161
Participants
  BPAR | 13 [1.51 to 1.81] | 13 [1.43 to 1.73] | 12 [1.61 to 1.91]
  Graft loss | 7 | 7 | 3
  Death | 7 | 4 | 9
  Lost to follow-up | 17 | 15 | 13
  Discontinuation due to adverse event | 10 | 8 | 4
  Therapy failure (composite endpoint) | 38 | 35 | 36

ADVERSE EVENTS:
Groups:
- CNI-free: CNI free regimen: comprising the following steps for switching treatment:
  Step 1 at BL2 + 1 day: Myfortic, Certican 1.5 mg, Sandimmun Optoral (50% of standard dose) and corticosteroids Step 2 at BL2 + 8 days: Myfortic, Certican 3 mg and corticosteroids
- CNI-low: CNI low regimen: comprising the following steps for switching treatment:
  Step 1 at BL2 + 1 day: Certican 1.5 mg, Sandimmun Optoral and corticosteroids Step 2 at BL2 + 8 days: Certican 1.5 mg, Sandimmun Optoral (low dose) and corticosteroids
Arm/Group | Standard Regimen | CNI-free | CNI-low
Serious Adverse Events (participants affected / at risk) | 87/165 | 91/171 | 85/161
Other Adverse Events (participants affected / at risk) | 121/165 | 134/171 | 133/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Regimen (N=165) | CNI-free (N=171) | CNI-low (N=161)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 1
BONE MARROW OEDEMA (Blood and lymphatic system disorders) | 0 | 1 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 4 | 1
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
POLYCYTHAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 2 | 0
ANGINA PECTORIS (Cardiac disorders) | 2 | 0 | 0
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2 | 1
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 1 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 0
CATARACT (Eye disorders) | 0 | 1 | 0
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 2 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 5 | 4
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0
NONINFECTIOUS PERITONITIS (Gastrointestinal disorders) | 0 | 1 | 0
RECTAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0
ATROPHY (General disorders) | 0 | 0 | 1
CHILLS (General disorders) | 1 | 0 | 0
DEVICE DISLOCATION (General disorders) | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0
IMPAIRED HEALING (General disorders) | 1 | 0 | 1
LOCALISED OEDEMA (General disorders) | 0 | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 3 | 4
SUDDEN CARDIAC DEATH (General disorders) | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 1 | 0
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 5 | 6 | 4
TRANSPLANT REJECTION (Immune system disorders) | 6 | 13 | 9
ANORECTAL INFECTION (Infections and infestations) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 2 | 1 | 0
BK VIRUS INFECTION (Infections and infestations) | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 2 | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0 | 2
CANDIDA INFECTION (Infections and infestations) | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 1 | 0 | 0
CYTOMEGALOVIRUS GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 6 | 1 | 4
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 0 | 1 | 0
DIABETIC GANGRENE (Infections and infestations) | 0 | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 0 | 1
ENCEPHALITIS (Infections and infestations) | 0 | 1 | 0
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 0 | 1 | 0
ESCHERICHIA INFECTION (Infections and infestations) | 0 | 1 | 0
FEBRILE INFECTION (Infections and infestations) | 1 | 0 | 2
GANGRENE (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 3 | 6 | 2
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 1 | 1 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1 | 2
GROIN ABSCESS (Infections and infestations) | 0 | 1 | 0
HAEMATOMA INFECTION (Infections and infestations) | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 2 | 1 | 1
INFECTION (Infections and infestations) | 4 | 1 | 1
INFLUENZA (Infections and infestations) | 0 | 0 | 1
KIDNEY INFECTION (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1 | 0
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 6 | 4
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 0 | 2 | 0
PNEUMONIA INFLUENZAL (Infections and infestations) | 0 | 1 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 1
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 | 0 | 2
PYELONEPHRITIS (Infections and infestations) | 1 | 1 | 0
PYONEPHROSIS (Infections and infestations) | 0 | 0 | 1
RENAL CYST INFECTION (Infections and infestations) | 1 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
SALPINGO-OOPHORITIS (Infections and infestations) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 1
SHUNT INFECTION (Infections and infestations) | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 15 | 12 | 7
UROSEPSIS (Infections and infestations) | 6 | 2 | 7
VARICELLA (Infections and infestations) | 1 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 1 | 1
WOUND INFECTION (Infections and infestations) | 1 | 1 | 0
ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
COMPLICATIONS OF TRANSPLANT SURGERY (Injury, poisoning and procedural complications) | 1 | 0 | 0
COMPLICATIONS OF TRANSPLANTED KIDNEY (Injury, poisoning and procedural complications) | 5 | 0 | 2
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
GRAFT LOSS (Injury, poisoning and procedural complications) | 0 | 2 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0 | 1
KIDNEY RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 | 0 | 0
RENAL LYMPHOCELE (Injury, poisoning and procedural complications) | 1 | 0 | 0
SEROMA (Injury, poisoning and procedural complications) | 1 | 0 | 0
SHUNT OCCLUSION (Injury, poisoning and procedural complications) | 0 | 1 | 1
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 2 | 0 | 1
TRANSPLANT DYSFUNCTION (Injury, poisoning and procedural complications) | 0 | 0 | 1
TRANSPLANT FAILURE (Injury, poisoning and procedural complications) | 3 | 5 | 3
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0
VENA CAVA INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 14 | 14 | 17
CARBOHYDRATE ANTIGEN 125 INCREASED (Investigations) | 0 | 0 | 1
CREATININE URINE INCREASED (Investigations) | 0 | 1 | 0
CYTOMEGALOVIRUS TEST (Investigations) | 2 | 0 | 0
CYTOMEGALOVIRUS TEST POSITIVE (Investigations) | 1 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1
IMMUNOSUPPRESSANT DRUG LEVEL INCREASED (Investigations) | 0 | 0 | 1
RED BLOOD CELL ACANTHOCYTES PRESENT (Investigations) | 1 | 0 | 0
WEIGHT INCREASED (Investigations) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
POST TRANSPLANT DISTAL LIMB SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
POST TRANSPLANT LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 2 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 1 | 0
POLYNEUROPATHY (Nervous system disorders) | 1 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 1
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 1 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1 | 2
GLOMERULOSCLEROSIS (Renal and urinary disorders) | 1 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 2 | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 1
KIDNEY FIBROSIS (Renal and urinary disorders) | 0 | 1 | 0
NEPHRECTASIA (Renal and urinary disorders) | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 1
NEPHROPATHY (Renal and urinary disorders) | 0 | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 0 | 3 | 1
REFLUX NEPHROPATHY (Renal and urinary disorders) | 1 | 0 | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 2 | 2 | 0
RENAL CYST RUPTURED (Renal and urinary disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 2 | 0 | 0
RENAL INFARCT (Renal and urinary disorders) | 1 | 0 | 0
RENAL TUBULAR ATROPHY (Renal and urinary disorders) | 0 | 1 | 0
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 | 0 | 2
URETERIC STENOSIS (Renal and urinary disorders) | 2 | 1 | 0
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 | 0 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 2 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 1
VESICOURETERIC REFLUX (Renal and urinary disorders) | 0 | 1 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 2 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0 | 0
ALVEOLITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
PLEURAL FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RESUSCITATION (Surgical and medical procedures) | 0 | 0 | 1
ARTERIAL HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0
ARTERIAL THROMBOSIS (Vascular disorders) | 1 | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 2 | 1
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 1
EMBOLISM (Vascular disorders) | 1 | 0 | 0
EMBOLISM ARTERIAL (Vascular disorders) | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 1 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0 | 0
LYMPHOCELE (Vascular disorders) | 2 | 1 | 4
LYMPHOEDEMA (Vascular disorders) | 0 | 0 | 1
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 0 | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 0 | 0 | 1
THROMBOSIS (Vascular disorders) | 0 | 0 | 3
VASCULITIS (Vascular disorders) | 0 | 1 | 0
VENOUS ANEURYSM (Vascular disorders) | 1 | 0 | 0
VENOUS OCCLUSION (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Regimen (N=165) | CNI-free (N=171) | CNI-low (N=161)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 14 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 22 | 26 | 18
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 | 33 | 14
DIARRHOEA (Gastrointestinal disorders) | 17 | 34 | 15
NAUSEA (Gastrointestinal disorders) | 5 | 8 | 9
OEDEMA (General disorders) | 15 | 14 | 22
OEDEMA PERIPHERAL (General disorders) | 9 | 17 | 28
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 12 | 8 | 4
NASOPHARYNGITIS (Infections and infestations) | 29 | 36 | 37
URINARY TRACT INFECTION (Infections and infestations) | 37 | 31 | 32
BLOOD CREATININE INCREASED (Investigations) | 14 | 11 | 12
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 4 | 8 | 18
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 4 | 6 | 11
HYPERURICAEMIA (Metabolism and nutrition disorders) | 9 | 3 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10 | 20 | 6
IRON DEFICIENCY (Metabolism and nutrition disorders) | 10 | 7 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 11 | 7
HEADACHE (Nervous system disorders) | 7 | 11 | 10
PROTEINURIA (Renal and urinary disorders) | 3 | 6 | 13
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 7
HYPERTENSION (Vascular disorders) | 10 | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.